CLINICAL TRIAL: NCT04240379
Title: Metacognition Assessment in Patient With Multiple Sclerosis
Acronym: METACOGSEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.146; 2019-A01278-49 (Other: ID RCB)
Record Dates: First submitted 2020-01-06; First posted 2020-01-27 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Multiple Sclerosis Functional Composite (MSFC); Metacognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assessed the level of consciousness of MS patients suffering of cognitive and motor disorders. Understanding the awareness of the disease is crucial to allow better management of these patients. It has been shown, for other neurological pathologies, that a lack of awareness of deficits leads to inefficient rehabilitation and a disorder of understanding the impact of deficits in daily activities. Metacognition could be altered with age, so we will include participants between 18 and 60 years old.

DETAILED DESCRIPTION:
Subject who have to do neurological assessement by the Multiple sclerosis Functional Composite (MSFC) will be enrolled.

The patient will estimate the time to undergo the test. This time will be compared to the time really make by the patient to realise test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Voluntary for participate to study

Exclusion Criteria:

* Neurological disease other than Multiple Sclerosis
* psychiatric disease, other than depressiveness
* illicit substance abuse
* Persons referred to in Articles L1121-5 to 8 of the French Public Health Code

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be proposed to subject :
  * Male or female with diagnosis of MS,
  * admitted in neurological unit for passing the MSFC (Multiple Sclerosis Functionnal Composite) test
  * who respect selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Metacognitive precision | Day 1
  Metacognitive precision based on Multiple Sclerosis Functional Composite (MSFC) score

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calabrese P. Neuropsychology of multiple sclerosis--an overview. J Neurol. 2006 Feb;253 Suppl 1:I10-5. doi: 10.1007/s00415-006-1103-1. PMID 16477479
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Result] Beatty WW, Monson N. Metamemory in multiple sclerosis. J Clin Exp Neuropsychol. 1991 Mar;13(2):309-27. doi: 10.1080/01688639108401046. PMID 1688342